CLINICAL TRIAL: NCT04273555
Title: Monitoring Early Response to Targeted Therapy in Stage IV Human Epidermal Growth Factor Receptor 2 Positive (HER2+) Breast Cancer Patients With Advanced Positron Emission Tomography (PET)/Magnetic Resonance Imaging (MRI)
Brief Title: Monitoring Early Response to Targeted Therapy in Stage IV HER2+ Breast Cancer Patients With Advanced PET/MR Imaging
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to recruit for this study.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Anna G. Sorace, Assistant Professor, Department of Radiology and Biomedical Engineering Director, The Small Animal Facility in the Advanced Medical Imaging Research Division, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R19-149; UAB (Other Grant/Funding Number: UAB Comprehansive Cancer Center and Department of Radiology)
Record Dates: First submitted 2020-01-30; First posted 2020-02-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: HER2-positive Breast Cancer
Keywords: FDG-PET; MRI; quantitative imaging
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- [18F]-Fluorodeoxyglucose (FDG) PET/ MRI (Experimental)
  Interventions: Drug: [18F]-FDG

INTERVENTIONS:
Drug: [18F]-FDG — [18F]-FDG will be injected prior to PET/MRI imaging up to three times over the course of six months.

SUMMARY:
The purpose of the study is to see if a new group of imaging tests can help identify response to stage IV HER2+ breast cancer before treatment.

DETAILED DESCRIPTION:
The purpose of this study is to see if a new group of imaging tests can help identify response to stage IV human epidermal growth factor receptor 2 positive (HER2+) breast cancer before and during treatment. This study will test a new method for monitoring treatment. The investigators will use [18F]-Fluorodeoxyglucose (FDG) positron emission tomography (PET)/magnetic resonance imaging (MRI) to look at previously diagnosed stage IV breast cancer and image up to three times during therapy. FDG is a non-natural amino acid with a radioactive tag that is used clinically for staging of disease. However, the role of FDG-PET/MRI for imaging response in breast cancer is not currently clear. PET/MRI is a new imaging technique that combines PET and MRI into a single study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years old and ≤ 75 years old
* Patients with HER2+ metastatic breast cancer
* HER2-positive breast cancer prospectively determined on the primary tumor by a local pathology laboratory and defined as immunohistochemistry (IHC) score of 3+ and/or positive by in situ hybridization (ISH) (defined by ISH ratio of ≥ 2.0 for the number of HER2 gene copies to the number of chromosome 17 copies). Only one positive result is required for eligibility
* Estrogen/progesterone receptor positive OR negative disease allowed
* Patients must have measurable disease in one metastatic lesion per RECIST v 1.1
* Stage IV HER2+ breast cancer patients eligible for a new therapeutic regimen that includes HER2-targeted treatment who are naïve to that regimen
* Estimated life expectancy of greater than six months

Exclusion Criteria:

* Children, less than 18 years of age, will be excluded from this study
* Metastatic breast cancer patients who are HER2 positive and have already started their current HER2-targeted therapy regimen for metastatic disease
* Patients who have not recovered from grade 2 or higher toxicities of prior therapy to the point that they would be appropriate for re-dosing will be ineligible for study treatment
* Patient is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit through 7 months after the last dose of study treatment
* Patient is considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease or active infection that requires systemic therapy. Specific examples include, but are not limited to, active, non-infectious pneumonitis; uncontrolled major seizure disorder; unstable spinal cord compression; superior vena cava syndrome; or any psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study (including obtaining informed consent).
* Patients found to have constitutionally present non-magnetic resonance (MR) compatible ferromagnetic materials
* Unable to lie still on the imaging table for one (1) hour
* Inability to receive gadolinium-based contrast agent
* Patients for whom a PET/MRI is technically not feasible (e.g. breast volume, obesity, > body mass index (BMI) 36)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Baseline measure of PET standardized uptake value (SUV). | Baseline imaging visit 1
  Compare baseline metrics from PET/MRI
Baseline measure of apparent diffusion coefficient (ADC) in mm2/sec from MRI. | Baseline imaging visit 1
  Compare baseline metrics from PET/MRI
Baseline measure of signal enhancement ratio (SER) from MRI. | Baseline imaging visit 1
  Compare baseline metrics from PET/MRI
Changes in SER from MRI | Baseline through 6 months
  Compare percent change of SER from imaging visit 3 to the baseline.
Changes in ADC from MRI | Baseline through 6 months
  Compare percent change of ADC (mm2/sec) from imaging visit 3 to the baseline.
Changes in SUV from PET | Baseline through 6 months
  Compare percent change of SUV from imaging visit 3 to the baseline.

SECONDARY OUTCOMES:
Follow-up | Baseline through 5 year follow-up
  Compare changes in imaging metrics to disease progression (defined as clinical progression of disease through increase in lesion size or increase in number of lesions).
Changes in ADC (mm2/sec) from MRI. | Baseline through 2 months
  Compare percent change from imaging visit 2 to the baseline.
Changes in SER from MRI. | Baseline through 2 months
  Compare percent change from imaging visit 2 to the baseline.
Changes in SUV from PET. | Baseline through 2 months
  Compare percent change from imaging visit 2 to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sorace, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No